CLINICAL TRIAL: NCT01999556
Title: LCI-HEM-SPEC-001: Tissue Collection for Familial Acute Myelogenous Leukemia Genetic Analysis
Brief Title: LCI-HEM-SPEC-001: Tissue Collection for Genetic Analysis of Acute Myelogenous Leukemia
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: LCI-HEM-SPEC-001; 00008179
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2022-04-21 (Actual); Status verified 2021-11

CONDITIONS: Leukemia, Myelogenous, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Specimen Collection
- Relative: Specimen Collection

SUMMARY:
The purpose of this study is to obtain high quality specimens for molecular studies for the identification and characterization of genetic mutations involved in the pathogenesis of familial myeloid malignancies. Specimens obtained will be de-identified, linked to basic clinical data, and sent to Washington University (Division of Oncology, St. Louis, MO) for molecular analyses. Some specimens sent to Washington University may also be used for quality control analyses.

DETAILED DESCRIPTION:
This is a specimen collection study for patients receiving standard of care treatment for AML. Specimens collected will be 1) bone marrow biopsy and aspiration, 2) peripheral blood, 3) skin punch biopsy, and 4) oral rinse. Collection of these specimens will be at timepoints determined by the patient's standard of care and their physician Investigator.

ELIGIBILITY:
Inclusion Criteria

* Patients must have a diagnosis of acute myelogenous leukemia.
* Family members of patients with acute myelogenous leukemia may be enrolled.
* Informed consent must be provided by the patient or his/her legal guardian in accord with the practices of Levine Cancer Institute and Atrium Health.

Exclusion Criteria

* Known infection with Hepatitis B or C, HTLV, or HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients must have a diagnosis of acute myelogenous leukemia. Family members of patients with acute myelogenous leukemia may be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2013-11; Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with the mutation for acute myelogenous leukemia. | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Druhan, PH.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States